CLINICAL TRIAL: NCT04347824
Title: Covid-19 Associated Nephritis as Early Predictor for Complicated Course of Disease
Brief Title: Predict Adverse Events by Covid-19 Nephritis
Status: Completed | Type: Observational
Sponsor: University Hospital Goettingen (Other)
Collaborators: Universitätsklinikum Hamburg-Eppendorf (Other); University Hospital, Aachen (Other); Transplantationszentrum Köln-Merheim (Other)
Responsible Party: Principal Investigator, Prof. Dr. O. Gross, Professor, University Hospital Goettingen
Other Study IDs: UMG_Co19-Nephritis
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- low risk: This group has a normal urine status on admission to hospital. Abnormal urine status is defined anuric OR as 2* or more of the following findings:
  1. urine osmolarity below normal values
  2. leukozyturia
  3. hematuria
  4. albuminuria/ proteinuria * if urine is positive for nitrite or bacteria, abnormal urine status is defined as 3 or more of the findings.
- intermediate risk: This group has an abnormal urine status on admission to hospital WITHOUT serum-albumin below 2.0 g/dl AND WITHOUT antithrombin III level below 70%.
- high risk: This group has an abnormal urine status on admission to hospital PLUS serum-albumin below 2.0 g/dl OR antithrombin III level below 70%.

SUMMARY:
This non-interventional, observational study retrospectively (and in parts prospectively) investigates, if a Covid-19 associated Nephritis, diagnosed by Urine-dipstick and further Urine-analyses on addmission, can help to predict later complications, adverse outcomes and later need for ICU-capacity in Covid-19 patients as well as can guide preventive strategies.

DETAILED DESCRIPTION:
Parameters predicting risks for Covid-19 patients are urgently sought. The current study investigates, if Covid-19 associated nephritis indicating systemic cappillary leak syndrome/severe nephrotic syndrome could be the major driver for complications, predictor for respiratory failure and later need for ICU, and death.

This study intends to generate an algorithm for University hospitals, which allows early detection of Covid-19 associated nephritis and to classify the risk for respiratory decompensation by quantification of severity of nephrotic syndrome.

The rationale of the observational study can be explained by the hypothesis that Covid-19 causes Nephritis: Podocytes express high levels of ACE2, which makes the glomerulus to a target for Covid-19. Other zoonoses, such as Hanta-virus, are a well described cause of nephrotic syndrome inducing cardiopulmonary syndrome. Life-threatening complications of severe nephrotic syndrome are well known as are preventive therapies.

Covid-19 ICU patients with nephritis have

1. pulmonary interstitial edema, possibly also due to capillary leak/ nephrotic syndrome;
2. immune-incompetence, due to renal loss of immunoglobulins;
3. circulatory insufficiency, due to hypalbuminemia (which might explain sudden deaths in the geriatric population);
4. less response to some medications caused by impaired plasma protein binding of drugs due to hypalbuminemia and renal loss;
5. thromboembolic events, due to antithrombin-deficiency (which might explain lethality in oligo-symptomatic young patients).

In conclusion, ACE2 in the respiratory tract is the gateway for Covid-19 for infection, however, the study postulates that Covid-19 associated nephritis and severe cappillary leak/nephrotic syndrome is a major driver of adverse outcome. If confirmed by others, these findings and algorithm would allow early prediction of later need for ICU-capacity, better allocation of patients for clinical trials, and preventive strategies focused on the nephrotic syndrome including treatment, which can save lives. Same might apply for risk-evaluation of outpatients.

ELIGIBILITY:
Inclusion Criteria:

1. approved Covid-19 diagnosis (by PCR or CT-scan);
2. urine status during hospital stay
3. Patient expressed willingness to participate in observational studies during hospital admission.

Exclusion Criteria:

1) Patient expressed unwillingness to participate in observational studies during hospital admission.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This observational study investigates the outcome of patients with approved Covid-19 diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 223 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Time to Disease-Aggravation | during first 10 days after admission to hospital
  Time (in days) from hospital admission to transferral to ICU (ICU level high) OR time (in days) from Hospital Admission to Death

SECONDARY OUTCOMES:
Complications | during first 10 days after admission to hospital
  Number of Complications are defined as
  1. Need of transferral to "ICU low" (ICU level 1)*
  2. Need of transferral to "ICU high" (ICU level 3)*
  3. Need of mechanical ventilation* OR
  4. Need for renal replacement therapy* OR
  5. Need of extracorporeal membrane oxygenation* OR
  6. Death * in the first 10 days after admission to hospital
Resources | during hospital stay, up to 2 months
  * Time on "ICU low" (in days),
  * Time on "ICU high" (in days),
  * Time on invasive mechanical ventilation (in days)
  * Time on extracorporeal membrane oxygenation (in days)
  * Time on renal replacement therapy (in days)
Blood-test | during hospital stay, up to 2 months
  * lowest serum-albumin
  * lowest antithrombin III

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Quesionnaires will be faxed to principal investigator and be analyzed by the department of medical statistics.

REFERENCES:
- [Background] Gross O, Moerer O, Weber M, Huber TB, Scheithauer S. COVID-19-associated nephritis: early warning for disease severity and complications? Lancet. 2020 May 16;395(10236):e87-e88. doi: 10.1016/S0140-6736(20)31041-2. Epub 2020 May 6. No abstract available. PMID 32423587
- [Background] Puelles VG, Lutgehetmann M, Lindenmeyer MT, Sperhake JP, Wong MN, Allweiss L, Chilla S, Heinemann A, Wanner N, Liu S, Braun F, Lu S, Pfefferle S, Schroder AS, Edler C, Gross O, Glatzel M, Wichmann D, Wiech T, Kluge S, Pueschel K, Aepfelbacher M, Huber TB. Multiorgan and Renal Tropism of SARS-CoV-2. N Engl J Med. 2020 Aug 6;383(6):590-592. doi: 10.1056/NEJMc2011400. Epub 2020 May 13. No abstract available. PMID 32402155
- [Derived] Gross O, Moerer O, Rauen T, Bockhaus J, Hoxha E, Jorres A, Kamm M, Elfanish A, Windisch W, Dreher M, Floege J, Kluge S, Schmidt-Lauber C, Turner JE, Huber S, Addo MM, Scheithauer S, Friede T, Braun GS, Huber TB, Blaschke S. Validation of a Prospective Urinalysis-Based Prediction Model for ICU Resources and Outcome of COVID-19 Disease: A Multicenter Cohort Study. J Clin Med. 2021 Jul 9;10(14):3049. doi: 10.3390/jcm10143049. PMID 34300217